CLINICAL TRIAL: NCT04369144
Title: Effect of Adding Continual Vertical Downward Correction to Dynamic Scapular Recognition Exercise on Scapular Dyskinesis and Shoulder Pain and Disability in Patients With Frozen Shoulder: a Randomized Controlled Trial
Brief Title: Adding Vertical Correction to Scapular Recognition on Patients With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Scapula recognition and taping
Record Dates: First submitted 2020-04-21; First posted 2020-04-30 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Double-blinded Randomized Controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The dynamic scapular recognition exercise + rigid taping with 50%-75% tension.
  Interventions: Other: Dynamic Scapular Recognition exercise
- Control (Placebo Comparator): The dynamic scapular recognition exercise + placebo taping
  Interventions: Other: Dynamic Scapular Recognition exercise

INTERVENTIONS:
Other: Dynamic Scapular Recognition exercise — The intervention group received continual vertical downward correction using a standardized rigid tape. A hypoallergenic tape (Hypafix; BSN Medical GmbH, Hamburg, Germany) was used with 50% to 75% tension. Two rigid tapes were applied; the first one is placed from just superior to the midpoint of the superior border of the scapula to the level of T12 and the second tapes were placed from just superior to the superior angle of the scapula to the level of T12. The level of T12 was used as the end of both taps to increase the lever arm of the applied force and to decrease the incidence of peeling off of the tape. No tape was applied from the lateral angle of the scapula because it might impair the upward rotation of the scapula. Both taps were performed after each session and removed immediately before the next session
  Other Names: Rigid Taping

SUMMARY:
OBJECTIVE: To study the effect of adding a continual vertical downward correction to dynamic scapular recognition exercise on scapular dyskinesis and shoulder pain and disability in patients with frozen shoulder.

Design: A double-blinded randomized controlled study Setting: Out-patient clinic Subjects: Sixty-seven subjects with unilateral frozen shoulder Interventions: Participants were distributed into two groups. The intervention group performed the dynamic scapular recognition exercise and continual vertical downward correction using rigid taping with 50%-75% tension. The control group performed a similar dynamic scapular recognition exercise using a wireless biofeedback system and placebo taping. A scapular dyskinesis test with caliper was utilized to measure scapular dyskinesis, a digital inclinometer was utilized to evaluate the scapular upward rotation and shoulder ROMs, and the Shoulder Pain and Disability Index (SPADI) was utilized to evaluate the shoulder pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* The existence of a unilateral frozen shoulder with incapability of the participant to raise the arm more than 100 degrees in the plane of the scapula.
* Aa restriction in both passive and active shoulder ROM
* The existence of pain that affects performing activities of daily living[19]

Exclusion Criteria:

* The presence of any shoulder problem contraindicated for performing exercises to the shoulder joint, such as active inflammatory disease, cancer, active infection, recent subluxations or dislocations, fractures, and surgeries nearby the shoulder region. Furthermore, the patient was excluded if he/she had no signs of scapular dyskinesis.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Scapular dyskinesis | 2 months
  Firstly, the patient was requested to place his/her upper limbs at his/her side with shoulders in mid-rotation and elbows straight. To better observation of scapular dyskinesis, this test was done with grasping dumbbells following the bodyweight, 1.4 kg (3 lb) for patients weighting lower than 68.1 kg (150 lb) and 2.3 kg (5 lb) for patients weighting 68.1 kg or higher. If any patient was unable to carry these predetermined weights, the weight was decreased by 0.5 kg(20). Then, the patient was instructed to instantaneously raise his arms overhead with thumbs-up as much as possible at a 3-second count and then lower arms back to the same starting position at a 3-second count.
Scapular Upward rotation | 2 months
  Digital inclinometers are reliable and validated tools in assessing the improvement in scapular upward rotation. During the test, the tested arm was preserved at 80 degrees of shoulder abduction. The upward rotation of the scapula was calculated as the angle formed between the line drained among lateral and medial parts of the spine of the scapula and the horizontal line drained parallel to the ground.
Shoulder Pain and disability index (SPADI) | 2 Months
  Before gathering information from the patients, a detailed clarification of the SPADI was provided to them. Then, patients were requested to represent the extent of their shoulder pain and disability by selecting one number on subscales from zero (no pain or disability) to ten (maximum pain and disability) for each item. The results of each subscale were summarized and converted to a score out of 100. The means of these two subscales were summarized to give a total score out of 100. The lower the final score, the better the shoulder pain, impairment or disability.

SECONDARY OUTCOMES:
Shoulder ROMs | 2 months
  The assessment of shoulder ROMs was performed by the similar digital inclinometer utilized for assessing scapular upward rotation. Digital inclinometers are reliable tools for assessing shoulder ROMs. For more precise assessment, the inclinometer was re-calibrated to zero degrees in advance of each measurement

CONTACTS AND LOCATIONS:
Locations (1):
- beni Suef University, Banī Suwayf, Egypt